CLINICAL TRIAL: NCT07347925
Title: Evaluating the Impact of Pre-Hospital Angiotensin Receptor-Neprilysin Inhibitor (ARNI) Therapy on Short-Term Clinical Outcomes in Heart Failure Patients With Reduced Ejection Fraction: A Comparative Study
Brief Title: Effect of Pre-Hospital ARNI Therapy on Short-Term Outcomes in HFrEF
Status: Recruiting | Type: Observational
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Mrwan Ayman Ahmed Eassa, MS Student, Clinical Pharmacy Department, Future University in Egypt, Future University in Egypt
Other Study IDs: REC-FPFUE-NO3/2025
Record Dates: First submitted 2025-12-15; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: Heart Failure; NYHA class; Sacubitril/Valsartan; Chronic kidney disease
MeSH Terms: conditions — Heart Failure; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Prehospital ARNI users
  Interventions: Other: Prehospital ARNI use
- Non-Prehospital ARNI users
  Interventions: Other: No prehospital ARNI use

INTERVENTIONS:
Other: Prehospital ARNI use — Participants who were using ARNI therapy before hospital admission
  Groups: Prehospital ARNI users
Other: No prehospital ARNI use — Participants who were not using ARNI therapy before hospital admission
  Groups: Non-Prehospital ARNI users

SUMMARY:
This study looks at people with heart failure who are admitted to the hospital. The goal of the study is to understand whether taking a heart failure medicine called angiotensin receptor-neprilysin inhibitor (ARNI) before hospital admission affects short-term health outcomes.

The study will compare two groups of participants: those who were already taking ARNI before coming to the hospital and those who were not. Information will be collected from medical records during the hospital stay, including heart-related events, kidney-related events, and how long participants stay in the hospital.

Some participants will also be followed for a short period after discharge. This study may help improve understanding of outcomes associated with ARNI use in people with heart failure in routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years, male or female EF <40%

Exclusion Criteria:

* EF>40% Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients with heart failure and reduced ejection fraction who are admitted to the cardiology wards at Mansoura University Hospital (MUH) during the study period. Participants include those who were already receiving ARNI therapy prior to hospital admission and those who were not, representing typical patients seen in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
In-hospital cardiac and renal events | 3 months

SECONDARY OUTCOMES:
NYHA classification | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university Hospital, Al Mansurah, Egypt